CLINICAL TRIAL: NCT02920164
Title: Auricular Acupuncture for Exam Anxiety in Medical Students: A Randomized Crossover Investigation
Brief Title: Auricular Acupuncture for Exam Anxiety in Medical Students
Acronym: AAAnx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BB 49/12
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auricular acupuncture (Active Comparator): Auricular acupuncture with indwelling fixed auricular acupuncture needles
  Interventions: Device: Auricular acupuncture
- Placebo acupuncture (Placebo Comparator): Placebo acupuncture with placebo fixed "needles"
  Interventions: Device: Placebo acupuncture
- Standard therapy (No Intervention): No intervention, just observation

INTERVENTIONS:
Device: Auricular acupuncture — Auricular acupuncture with indwelling permanent needles
  Arms: Auricular acupuncture
Device: Placebo acupuncture — Placebo acupuncture with placebo needles
  Arms: Placebo acupuncture

SUMMARY:
Title of the study: Auricular acupuncture (AA) for pre-exam anxiety: A blinded randomized crossover study on healthy volunteers

Study period: 04/2012 - 07/2012

Institution: Department of Anesthesiology and Intensive Care Medicine University Medicine of Greifswald

Aim of the study: To investigate the anxiolytic effect of auricular acupuncture (AA) in comparison to placebo acupuncture and no intervention during oral exams in anatomy at the University of Greifswald

Design: Prospective blinded randomized crossover trial

Intervention:

1. AA using indwelling fixed needles, retained 24 h in situ
2. AA using placebo needles

Number of volunteers: N = 40

Outcome measures: Anxiety level, Heart rate, blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Medical students at the University of Greifswald
2. Going to take part in oral exams of human anatomy
3. Participants without previous anxiolytic medication
4. Participants without any experiences with acupuncture
5. Patients who have given written informed consent

Exclusion Criteria:

1. Local auricular skin infection
2. Pregnant or lactating women
3. Participants with prosthetic or damaged cardiac valves, intracardiac and intravascular shunts, hypertrophic cardiomyopathy and mitral valve prolapse (risk of bacterial endocarditis according to guidelines of AHA)
4. Participants who are unable to understand the consent form
5. History of psychiatric disease, alcohol and drug abuse

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Intensity of anxiety | 2 days
  State-Trait-Anxiety Inventory

SECONDARY OUTCOMES:
heart rate | 1 day
blood pressure | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Taras Usichenko, MD, PhD, Study Chair — University Medicine of Greifswald
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided